CLINICAL TRIAL: NCT01189695
Title: A Randomized Controlled Study Compares the 48 Weeks Results of HIV-1 RNA Between Ritonavir-boosted Lopinavir Monotherapy and Ritonavir-boosted Lopinavir + Optimized Background Regimens in HIV-1 Infected Patients Who Have HIV-1 RNA <50 Copies/ml More Than 6 Months While Receiving Salvage PI-based Regimen and Previously Failed NNRTI-based Regimen
Brief Title: Maintenance Boosted Lopinavir Monotherapy Following Salvage Protease-inhibitor (PI) Based Regimen in HIV With Non-nucleoside Reverse Transcriptase Inhibitors (NNRTI) Based Regimen Failure
Acronym: BIDI-MONO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bamrasnaradura Infectious Diseases Institute (Other Government)
Collaborators: Department of Disease Control, Thailand (Unknown)
Responsible Party: Principal Investigator, Krittaecho Siripassorn, Dr, Bamrasnaradura Infectious Diseases Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIDI-MONO
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: HIV; AIDS; Lopinavir; Treatment Failure
Keywords: HIV or AIDS; Lopinavir; Ritonavir; Anti-Retroviral Agents; treatment failure; treatment experienced; NNRTI failure; monotherapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Boosted lopinavir monotherapy (Experimental)
  Interventions: Drug: Ritonavir-boosted lopinavir
- boosted lopinavir + optimized background regimens (OBRs) (Active Comparator)
  Interventions: Drug: Ritonavir-boosted lopinavir; Drug: optimized background regimens (OBRs)

INTERVENTIONS:
Drug: Ritonavir-boosted lopinavir — Lopinavir/ritonavir 200/50 mg every 12 hours
Drug: optimized background regimens (OBRs) — Optimized background regimens such as NRTIs, etravirine or raltegravir
  Arms: boosted lopinavir + optimized background regimens (OBRs)

SUMMARY:
The objective of this study is to determine efficacy of ritonavir-boosted lopinavir monotherapy as a maintenance regimen in HIV-1-infected patients who previously failed Non-nucleoside reverse transcriptase inhibitors (NNRTI) based regimens and currently received salvage protease-inhibitor (PI) based regimens.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* documented HIV infection
* previously failed to NNRTI-based regimens
* no history of failing PI-based regimens
* receiving ritonavir-boosted PI + OBRs(such as NRITs, etravirine, raltegravir)
* having HIV-1 RNA <50 copies/ml for at least prior 6 months

Exclusion Criteria:

* Pregnant or breastfeeding woman
* HBV co-infection that had to treated with TDF, FTC or 3TC
* had to received medications known to have potential significant drug interaction with LPV/r
* life expectancy less than 6 months
* serious systemic diseases such as liver cirrhosis Child-Pugh B/C, ESRD, malignancy
* hemoglobin <8 g/dl, platelet <50,000/mm3, AST or ALT >3 ULN, estimated creatinine clearance <50 mL/min

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Time to virological failure | 48 weeks
  virological failure was defined as having two consecutive results of HIV-1 RNA >400 copies/ml in time separated by 4 weeks

SECONDARY OUTCOMES:
Proportion of patients with virological suppression | 48 weeks
  virological suppression defined as having HIV-1 RNA <40 copies/ml
Proportion of patients with virological failure | 48 week
  virological failure was defined as having two consecutive results of HIV-1 RNA >400 copies/ml in time separated by 4 weeks
Time to loss of virological response (TLOVR) | 48 weeks
  TLOVR was defined as time between randomization and the last value that HIV-1 RNA <40 copies/ml in a patient who initially suppressed HIV-1 RNA but subsequently demonstrated virologic rebound (two consecutive HIV-1 RNA >40 copies/ml)
Change of CD4 cells count | 48 weeks
  Change of CD4 cells count from start of study to Week 48
Adverse events | 48 weeks
  any grade 3 or grade 4 adverse events according to DAIDS AE grading table

CONTACTS AND LOCATIONS:
Overall Officials: Krittaecho Siripassorn, MD, Principal Investigator — Bamrasnaradura Infectious Diseases Institute
Locations (1):
- Bamrasnaradura Infectious Diseases Institute, Nonthaburi, Thailand